CLINICAL TRIAL: NCT04446754
Title: The Association Between TCF7L2 rs7903146, Diet and Type 2 Diabetes Mellitus Risk
Brief Title: The Genetic Effects of rs7903146 and Dietary Intake on Type 2 Diabetes Mellitus Risk in a Healthy Population
Status: Completed | Type: Observational
Sponsor: St Mary's University College (Other)
Responsible Party: Sponsor
Other Study IDs: SMEC_2018-19_034
Record Dates: First submitted 2020-06-19; First posted 2020-06-25 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Health Behavior; Blood Glucose, High; Diet Habit; Genetic Predisposition
MeSH Terms: conditions — Health Behavior; Feeding Behavior; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva and blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study investigates the association of genetic effects of rs7903146 and dietary intake on type 2 Diabetes Mellitus (T2DM) risk in a healthy population. T2DM risk was assessed through glycated haemoglobin (HbA1c) concentration in 73 subjects. Dietary intake was assessed using a validated food frequency questionnaire (FFQ).

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) is a global epidemic linked to 1.6 million deaths in 2016. Diet, lifestyle and environment contribute significantly to T2DM-risk. Genome-wide association studies identify the transcription factor 7-like 2 (TCF7L2) rs7903146 (C/T) gene as one of the most important associated with T2DM-risk. The T-allele is associated with a two-fold increase in relative risk of T2DM across different populations. However, most studies associating genetic effects of dietary intake on rs7903146 and T2DM-risk utilised volatile instantaneous measures of glucose(5) and focussed on individual macronutrients. Understanding the association of rs7903146 and overall macronutrient intake using a stable blood homeostasis marker may provide a fuller insight into T2DM-risk.

The study included data for all variables (participant characteristics: sex (female/male), age (years), height (cm), weight (kg), body mass index (BMI) (kg/m2), body fat percentage (%), fat mass (kg), lean mass (kg), waist/hip (ratio), dietary intake, HbA1c (mmol/mol and %) and physical activity (hours/week). All data was collected at St Mary's University between April to July 2019. Participants was genotyped and allocated into two groups: major allele (C) homozygote versus minor allele (T) homozygote plus heterozygote. T2DM-risk was assessed through their value of HbA1c and participants were classified as follows: normal (<42mmol/mol/ <6.0%), pre-diabetic (42 to 47 mmol/mol/ 6.0% to 6.4%), diabetes (48mmol/mol /6.5% or over).

ELIGIBILITY:
Inclusion criteria: Eligibility criteria required healthy adults free from metabolic condition and free from medication affecting glycated haemoglobin levels.

Exclusion criteria: Individuals with HbA1c levels ≥48 mmol/mol or ≥6.5% were excluded due to a classification as T2DM (WHO, 2011).

Ages: 18 Years to 64 Years | Sex: All
Age Groups: Adult
Study Population: Male-female age between 18 to 64.9 years old
Sampling Method: Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-10-02 (Actual)

PRIMARY OUTCOMES:
DNA | 3 months
  salivary (1-ml) DNA for genotype TCF7L2 gene (rs7903146 SNP)
Hba1c | 3 months
  capillary blood collected (via the ears or fingers) using a Microvette CB Lithium Heparin tube (SARSTEDT AG & C0., Nümbrecht, Germany)
Diet intake | 3 months
  Dietary intake estimated using The European Prospective Investigation into Cancer and Nutrition (EPIC)-Norfolk (food frequency questionnaire)

SECONDARY OUTCOMES:
Body weight | 3 months
  Body weight in kg measured by bioelectrical impedance analysis using a 0.5kg clothing offset
Waist | 3 months
  Waist measurement was taken midway between iliac crest and lowest rib
Hip | 3 months
  Hip circumference was measured over the greater trochanters at their widest point (nearest 0.1cm)
Height | 3 months
  Subject height was recorded to the nearest 0.1-cm via stadiometer
Physical activity | 3 months
  Assessed through Physical Activity Readiness Questionnaire (PAR-Q)
Fat mass | 3 months
  Measured in kg and percentage (%) measured by bioelectrical impedance analysis
Lean mass | 3 months
  Measured in kg and percentage (%) measured by bioelectrical impedance analysis

CONTACTS AND LOCATIONS:
Locations (1):
- St Marys University, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Podboi ICR, Stephenson S, Pilic L, Graham CA, King A, Mavrommatis Y. Dietary Intake and TCF7L2 rs7903146 T Allele Are Associated with Elevated Blood Glucose Levels in Healthy Individuals. Lifestyle Genom. 2021;14(4):117-123. doi: 10.1159/000518523. Epub 2021 Aug 12. PMID 34515148